CLINICAL TRIAL: NCT04275024
Title: Efficacy and Safety of AD-MSCs Plus Calpocitriol Ointment and PSORI-CM01 Granule in Patients With Moderate to Severe Psoriasis
Brief Title: Efficacy and Safety of AD-MSCs Plus Calpocitriol Ointment and PSORI-CM01 Granule in Psoriasis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chuanjian Lu, Professor, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2016-05-02
Record Dates: First submitted 2020-02-16; First posted 2020-02-19 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Mesenchymal Stromal Cells; Psoriasis; Drug Effect; Drug Toxicity
MeSH Terms: conditions — Psoriasis; Drug-Related Side Effects and Adverse Reactions | interventions — calcipotriene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): AD-MSCs: adipose-derived multipotent mesenchymal stem cells intravenous injection at a dose of 2 million cells/kg of body weight at week 0, week 2, week 4, week 6, week 8 with a duration for treatment for 12 weeks.
  The basic treatment is oral PSORI-CM01 Granule plus calcipotriol ointment (Dovonex;LEO Laboratories Ltd, Ireland) for topical use twice daily for 12 weeks.
  Interventions: Drug: Calcipotriol ointment; Drug: PSORI-CM01 Granule; Biological: adipose-derived multipotent mesenchymal stem cells

INTERVENTIONS:
Drug: Calcipotriol ointment — The topical treatment in the study was calcipotriol ointment(Dovonex;LEO Laboratories Ltd, Ireland) twice daily for 12 weeks.
  Other Names: Dovonex
Drug: PSORI-CM01 Granule — PSORI-CM01#YXBCM01# granule 5.5g os once a day for 12weeks.
  Other Names: Chinese Herbal Medicine
Biological: adipose-derived multipotent mesenchymal stem cells — AD-MSCs(adipose-derived multipotent mesenchymal stem cells) were infused intravenously at a dose of 2 million cells/kg

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Adipose derived Mesenchymal Stem Cells (AD-MSCs) plus Calpocitriol Ointment and PSORI-CM01 Granule with moderate to severe psoriasis. Any adverse events related to AD-MSCs infusion will be monitored.The primary outcome is the reduction rate of PASI(Psoriasis Area and Severity Index) and treatment response will be computed from PASI before and after treatment.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of Adipose derived Mesenchymal Stem Cells (AD-MSCs) plus Calpocitriol Ointment and PSORI-CM01 Granule with moderate to severe psoriasis. Any adverse events related to AD-MSCs infusion will be monitored.The primary outcome is the reduction rate of PASI(Psoriasis Area and Severity Index) and treatment response will be computed from PASI before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. moderate to severe psoriasis vulgaris ( PASI > 10 or BSA >10%)
2. 18 to 65 years old
3. written/signed informed consent

Exclusion Criteria:

1. guttate psoriasis, inverse psoriasis or exclusively associated with the face
2. Acute progressive psoriasis, and erythroderma tendency
3. current (or within 1 year) pregnancy or lactation
4. current significant anxiety or depression with the Self-rating Anxiety Scale (SAS) > 50 or the Self-rating Depression Scale (SDS) > 53, or with other psychiatric disorders
5. With history of primary cardiovascular, respiratory, digestive, urinary, endocrinologic and hematologic diseases, which can't be controlled through ordinary treatments. Those who with malignant diseases, infections, electrolyte imbalance, acid-base disturbance. Patients with clinical test results listed below: abnormal serum calcium level ( Ca2+ > 2.9 mmol/L or < 2 mmol/L);AST or ALT 2 times more than normal upper limit; Creatinine and cystatin C more than normal upper limit; Hemoglobin elevates 20g/L more than normal upper limit,or hemoglobin reduction to anemia; Platelet count less than 75.0*10^9/L; White blood cell less than 3.0*10^9/L; Or any other abnormal laboratory test results, assessed by investigators, that are not suitable for this clinical study
6. Patients with malignant tumors, or when they were enrolled with abnormal tumor markers or with other organ dysfunction
7. allergy to anything else ever before;
8. current registration in other clinical trials or participation within a month;
9. topical treatments (i.e. corticosteroids or retinoic acid or Vitamin D analogs ) within 2 weeks; systemic therapy or phototherapy (ultraviolet radiation B,UVB) and psoralen combined with ultraviolet A (PUVA) within 4 weeks; biological therapy within 12 weeks;
10. medical conditions assessed by investigators, that are not suitable for this clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
PASI score improvement rate | 12 weeks (plus or minus 3 days) after treatment
  PASI score improvement rate = (PASI score before intervention - PASI score after intervention)/PASI score before intervention ×100%

SECONDARY OUTCOMES:
PASI(Psoriasis Area and Severity Index) | 12 weeks (plus or minus 3 days) after treatment
  The improvement in PASI score from baseline after treatment
PASI-50 | 12 weeks (plus or minus 3 days) after treatment
  The proportion of patients who achieve at least 50% improvement in PASI score from baseline
PASI-75 | 12 weeks (plus or minus 3 days) after treatment
  The proportion of patients who achieve at least 75% improvement in PASI score from baseline
Pruritus Scores on the Visual Analogue Scale | 12 weeks (plus or minus 3 days) after treatment
  Pruritus was assessed using the Visual Analogue Scales; The Scale scores ranged from 0-10. The higer the scores were, the more itching the patient suffered
BSA | 12 weeks (plus or minus 3 days) after treatment
  the Body Surface Area
DLQI(Dermatology Life Quality Index) | 12 weeks (plus or minus 3 days) after treatment
  the Dermatology Life Quality Index

CONTACTS AND LOCATIONS:
Overall Officials: Chuanjian Lu, PhD, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong, China